CLINICAL TRIAL: NCT05838443
Title: Pragmatic Randomized Controlled Trial Evaluating Efficacy of Presurgical Provider-directed Behavioral and Self-directed Mindfulness Interventions in Pediatric Patients Undergoing Major Elective Surgical Procedures on Postoperative Pain Outcomes
Brief Title: Mindfulness Surgical Pain Outcomes
Acronym: MNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The Society for Pediatric Anesthesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0008
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Post Surgical Pain; Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-directed mindfulness (Active Comparator)
  Interventions: Other: Self-directed mindfulness utilizing a multi-sensor EEG-supported device with neurofeedback-assisted and technology-supported meditation
- Provider-directed mindfulness (Active Comparator)
  Interventions: Other: Provider-directed mindfulness
- Conventional care (Other): Control Comparator
  Interventions: Other: Conventional Care

INTERVENTIONS:
Other: Self-directed mindfulness utilizing a multi-sensor EEG-supported device with neurofeedback-assisted and technology-supported meditation — Neurofeedback-assisted, technology-supported mindfulness via EEG-supported device delivered individually without the need for a facilitator or travel to training site. The device allows noninvasive neural activity recording from frontal and posterior brain regions. A dedicated smartphone application uses the EEG data to provide real-time adaptive feedback-modulating natural sounds to prompt user awareness of mind-wandering and intentional return to present experience. A smartphone app will guide patients through attention and focus on breath exercises. Patients will hear their distracted mind as the wind. Wind becomes stronger if their mind wanders, prompting patient's awareness of their wandering mind and guiding the patient back to focusing on their breath without judgment of how they are doing. Patients will be asked to practice mindfulness using the device for 20 minutes per day for 4 sessions prior to surgery.
  Arms: Self-directed mindfulness
Other: Provider-directed mindfulness — Patients will receive mental health support by a licensed social work provider who is trained in mindfulness through four 20-minute telehealth sessions. Patients will be taught cognitive behavioral therapy (CBT) techniques to reduce pain catastrophizing and increase coping efficacy, the clinician will review patient's current sleep routine and teach concepts and strategies to improve sleep. Patients will be guided through mindfulness and meditation exercises to improve pain and mood coping. Mindfulness-based instructions takes patients through quieting their mind by focusing on breath, expanding focus (i.e., "at the tip of their nose" "full flow of the breath"), with emphasis on acknowledgement of arising thoughts/emotions without judgement or emotional reaction, and return attention back to breath sensation. Principles of CBT and mindfulness will be reiterated at subsequent sessions.
  Arms: Provider-directed mindfulness
Other: Conventional Care — Control group, as defined by our institution's standard preoperative care for given procedure, which does not include psychological preparation.
  Arms: Conventional care

SUMMARY:
This will be a prospective randomized study to evaluate novel, clinically feasible, easily deliverable, pragmatic ways of preemptively modifying known CPSP and behavioral risk factors for acute to chronic pain transitions in adolescents before surgery. In addition, it will provide mechanistic insights and build a strong foundation for future large scale interventional studies that can impact outcomes positively in children undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 10-18 years
2. English speaking
3. Ability to provide assent/consent/parent permission
4. Scheduled to undergo elective major musculoskeletal surgeries including spine fusion (idiopathic scoliosis only), abdominal surgeries, thoracic surgery including pectus repair, and major orthopedic joint surgeries.

Exclusion Criteria:

1. Previous exposure to psychological interventions
2. Surgery within 1 year
3. Developmental delay
4. Chronic opioid use within 6 months prior to surgery
5. Severe systemic disease

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Functional Disability Index (FDI) | Baseline pre-intervention, post-operatively at 1 week, 2 weeks and 4 months.
  15-item survey that assesses the extent to which children experience difficulties in completing specific tasks (for example, walking to the bathroom, eating regular meals, and being at school all day).

SECONDARY OUTCOMES:
Child and Adolescent Mindfulness Measure (CAMM) | Baseline pre-intervention, post-operatively at 1 week, 2 weeks and 3-4 months.
  10-item to assess 3 out of 4 facets of mindfulness: observing, acting with awareness and accepting without judgement. Scale is 0-40 with reverse scoring 0-4, 0 being never true, 4 being always true. Higher scores correspond to higher levels of mindfulness.
Child Anxiety Sensitivity Index (CASI) | Baseline pre-intervention, post-operatively at 1 week, 2 weeks and 3-4 months.
  18-item self-report tool designed to measure symptoms of anxiety in children and adolescents, with total scores ranging from 18-54. The CASI has demonstrated high internal consistency in both clinical and nonclinical samples (aged 8-15.8 years), good test-retest reliability and good construct validity.
Electronic Pain Diary and PainDETECT | Baseline pre-intervention, post-operatively at 1 week, 2 weeks and 3-4 months.
  Numerical rating pain scores of average pain intensity based on electronic pain ratings for one week, activity and sleep, using free phone application ("Manage my Pain" for Android and "Pain Diary" for iPhone users). PainDETECT assesses pain nature, with high sensitivity, specificity and positive predictive accuracy in pain conditions.
Perioperative Opioid use | Postoperative inpatient (if applicable), 1 week, 2 weeks and 3-4 months postoperatively.
  Opioid use over 4 months (total morphine equivalent dose standardized by weight). Post-operative opioid use will be obtained from electronic medical record if patient was admitted, as well as by patient/family report.
PROMIS pain interference-short form | Baseline pre-intervention, post-operatively at 1 week, 2 weeks and 3-4 months.
  8 items assessing how pain interferes with daily activities such as ambulating and doing school work. Total score range 8-40.
Pain Coping Efficacy | Baseline pre-intervention, post-operatively at 1 week, 2 weeks and 3-4 months
  Evaluate pain coping as a mediator of association of the intervention with long-term functional and pain outcomes utilizing a 3-item subsurvey from a 39-item self-report questionnaire (PHQ pain coping questionnaire) to assess pain coping strategies and pain coping efficacy in children.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio, United States